CLINICAL TRIAL: NCT03197753
Title: Postoperative Discomfort and Emergence Delirium In Children Receiving Dental Treatment Under General Anesthesia: Comparison Of Nasal Tracheal Intubation and Laryngeal Mask Airway
Brief Title: Postoperative Discomfort After Dental General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SULTAN KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/011
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain
Keywords: laryngeal mask airway; nasotracheal intubation; dental treatment
MeSH Terms: conditions — Pain, Postoperative | interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngeal mask airway (Experimental): Laryngeal mask airway insertion
  Interventions: Device: Laryngeal mask airway
- Nasotracheal intubation (Active Comparator): Nasotracheal tube insertion
  Interventions: Device: Nasotracheal intubation

INTERVENTIONS:
Device: Laryngeal mask airway — Laryngeal mask airway
  Arms: Laryngeal mask airway
Device: Nasotracheal intubation — Nasotracheal intubation
  Arms: Nasotracheal intubation

SUMMARY:
The aim of this prospective, randomised, controlled clinical trial was to compare immediate postoperative discomfort, emergence delirium and recovery time of the patients intubated using either laryngeal mask airway or nasotracheal intubation.

DETAILED DESCRIPTION:
A total of 70 children aged 3 to 7 years received full mouth dental rehabilitation under general anesthesia. Children were randomly grouped into Laryngeal mask airway (LMA) group (n=35) and nasotracheal intubation (NTI) groups (n=35). In LMA group LMA was inserted after anesthesia induction using 8% sevoflurane. In NTI group rocuronium and remifentanil were given intravenously during %8 sevoflurane induction and the patients were intubated by a nasotracheal tube. After completion of the dental treatments patients were transferred to the post anesthesia care unit (PACU). Duration of dental operation ,duration of anesthesia, recovery time, postoperative discomfort, emergence delirium, pediatric dentist's access were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-7 years,
* ASA I and II
* Lack of chairside cooperation for dental treatment in clinical setting.

Exclusion Criteria:

* A history of of anticipated difficult entubation ,
* Patient with pharyngeal pathology patients with known pulmonory or cardiovascular disease,
* When the expected dental procedure was more than two hours
* Mental retardation and those whose parents did not consent to their participation in the study.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Postoperative discomfort | Postoperative 1 hour
  Sore throat

CONTACTS AND LOCATIONS:
Overall Officials: Sultan KELES, Dr., Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Sultan Keles, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hung WT, Chen CC, Chau MY, Tsai WY. Effect of reinforced laryngeal mask airway or endotracheal intubation anesthesia on adverse events: quality of life issues for dental patients requiring general sedation. Spec Care Dentist. 2005 Jul-Aug;25(4):188-92. doi: 10.1111/j.1754-4505.2005.tb01648.x. PMID 16295223
- [Background] Zhao N, Deng F, Yu C. Anesthesia for pediatric day-case dental surgery: a study comparing the classic laryngeal mask airway with nasal trachea intubation. J Craniofac Surg. 2014 May;25(3):e245-8. doi: 10.1097/SCS.0000000000000547. PMID 24820727